CLINICAL TRIAL: NCT05873699
Title: Pilot Study Using Hyperpolarized 13C-Pyruvate Magnetic Resonance Spectroscopic Imaging in Patients With Pancreatic Cysts Undergoing Surgical Resection
Brief Title: Study Using Hyperpolarized 13C-Pyruvate Magnetic Resonance Spectroscopic Imaging in Patients With Pancreatic Cysts Undergoing Surgical Resection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-0854; NCI-2023-04096 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hyperpolarized 13C-Pyruvate Magnetic Resonance Spectroscopic Imaging (Experimental): Participants will have the HP-MR scan within the 4 weeks before your scheduled surgery.
  Hyperpolarized C-Pyruvate will be injected by vein during the scan. Your vital signs (temperature, blood pressure, heart rate and respiration [breathing]) will be monitored during the scan. The estimated time of the scan is a couple of minutes, but you may be in the room of the MRI for up to 30 minutes for preparation. The entire process of obtaining the MRI (and possible blood draw) may be up to half of a work day (not including your personal travel time).
  Interventions: Drug: Hyperpolarized 13-C-pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13-C-pyruvate — Given by Injection

SUMMARY:
To learn if Hyperpolarized C-Pyruvate Magnetic Resonance (HP-MR) Spectroscopic Imaging can help doctors detect low-risk (benign) and high-risk (malignant) cysts.

DETAILED DESCRIPTION:
Primary Objectives:

To explore the use of HP-MR in patients with cystic lesions of the pancreas undergoing surgical resection. Patients will undergo HP-MR prior to surgical resection (or cyst wall biopsy) and kpl values will be determined to evaluate metabolic activity. Pathology will then determine whether the cyst was of benign/low risk or malignant/high risk nature. The ability for increased kpl to detect an invasive carcinoma will be explored by estimating the association between lesions' kpl values and lesions' pathological results.

Secondary Objectives:

* A kpl inflection point, or threshold, will then be explored to estimate the association with malignant/high risk cyst. This threshold value would then undergo further validation in future studies to calculate the sensitivity and specificity of this value.
* Correlate HP-MR findings to tissue metabolomics (ex vivo): In all patients who undergo surgical resection, a small surgical sample will be supplied for ex vivo metabolomics. NMR metabolomics will be used to measure lactate, creatine, choline, phosphocholine, glycerophosphocholine, and alanine within the tissue sample. The highest lactate levels should be found in the most aggressive tumors, which also should correlate to high kpl.
* Correlate HP-MR findings to blood and cyst fluid biomarkers: Blood samples taken prior to surgical resection will be analyzed for CA19-9 and CEA. If the patient has a cystic fluid aspiration prior to surgical resection, then CA19-9, amylase and CEA will also be measured in these samples. These biomarkers will be compared to findings from HP-MR and pathologic results.
* Correlate HP-MR findings to immunohistochemical staining for LDH-A and HIF-1α: Tissue taken from pathology samples for metabolomics will also undergo immunohistochemical staining for LDH-A and HIF-1α.
* Correlate gut and tissue microbiome with HP-MR findings: Microbiome studies may be performed under the auspice of another protocol but could be analyzed under this protocol in relation to HP-MR findings. PA 16-0911 allows for the collection of stool in patients with cysts of the pancreas for gut microbiome investigation in relation to the development of pancreatic cancer.
* To explore the safety and tolerability of HP-MR in patients with cystic lesions of the pancreas undergoing surgical resection or cyst wall biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old. Patients under 18 are excluded due to their potential inability to understand and consent independently to the methods required for the study drug use and its potential risks and benefits.
* Patients with pancreatic cyst/s
* Patients who will undergo surgical resection (or cyst wall biopsy) of pancreatic cysts
* Patients able to understand and willing to sign a written informed consent document
* Both English-speaking and non-English-speaking patients are eligible for participation

Exclusion Criteria:

* Contraindication to MRI
* Electrically, magnetically, or mechanically activated implants that would preclude MRI
* Allergy to Gadavist IV contrast
* History of cardiac arrhythmias
* Pregnancy or breastfeeding women
* Women of child-bearing age that are sexually active and not using birth control
* Cognitively impaired individuals
* Weight above 260 pounds (lbs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Florencia McAllister, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org